CLINICAL TRIAL: NCT05180019
Title: Self Monitoring Device (SMD) for Trasvaginal Ultrasound in Reproduction
Brief Title: Self Monitoring Device Fortrasvaginal Ultrasound in Reproduction
Acronym: AUTOECOSMD
Status: Completed | Type: Observational
Sponsor: IVI Bilbao (Other)
Responsible Party: Sponsor
Other Study IDs: 2009-BIO-057-PR
Record Dates: First submitted 2021-12-17; First posted 2022-01-06 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Self-Evaluation
Keywords: Trasvaginal ultrasound 3D; Self-Monitoring Device; Pelvic ultrasound volume; risks; Trasvaginal ultrasound 2D

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient COS IVI Bilbao: Patients will come to the IVIRMA Bilbao clinic to start their respective ART cycles (vitrification, IVF/ICSI, donors) following usual clinical practice.
  Interventions: Device: SMD ( Self Monitoring Device)

INTERVENTIONS:
Device: SMD ( Self Monitoring Device) — Automated 3D ultrasound based follicullometry with SMD self-performed by the patient.
  Other Names: No names

SUMMARY:
Serial ultrasound (US) examinations are performed to assess the number and size of follicles during controlled ovarian stimulation (COS). Ovarian folliculometry during COS is the most frequent ultrasound procedure daily performed, an also a highly time consuming and reiterative process.

However, it has been shown that manual measurement of follicles with 2D US is often inaccurate and subject to significant intra- and interobserver variability

In addition, a follicle is a three-dimensional (3D) structure and its volume is the most accurate measure of its size. Therefore, 3D transvaginal ultrasound in gynaecology and reproductive medicine has supposed a great advance, because it makes possible to obtain ovarian volumes during controlled ovarian stimulation

DETAILED DESCRIPTION:
At each visit, IVIRMA Bilbao doctors (MF, CF) will perform routine folliculometry to the patients (standard 2D manual ultrasound) to control the ovarian stimulation. In this exam, follicles will be counted and measured (mean diameter) in millimeters, as usual clinical practice,

After the standard folliculometry, will request the patient for self-performing scan (3Dultrasound)

After each patient self-capture, IVIRMA Bilbao gynaecologists will check the saved volume (3D multiplanar mode) using ITKSnap viewer to ensure the correct acquisition saving (complete ovaries and uterus captured inside without artifacts) in order to compare 2D ultrasound (clinical reference) for number and mean follicle diameter estimations, with 3D multiplanar ultrasound (obtained with SMD) GMDN (Global Medical Device Nomenclature): 40761

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent form dated and signed
2. Female, aged 18 years or above
3. Patient undergoing COS for IVF/ICSI, oocyte vitrification or oocyte donation cycles in IVIRMA Bilbao clinic
4. Willing to comply with all study requirements

Exclusion Criteria:

1. Simultaneous participation in another clinical study that, at researcher's criteria, could interfere with the results of this study.
2. Any significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The target population includes any women who wants to carry out a COS for IVF/ICSI, oocyte donor or oocyte vitrification treatment
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2022-02-09 (Actual); Primary Completion 2023-05-08 (Actual); Study Completion 2023-05-08 (Actual)

PRIMARY OUTCOMES:
SMD validation for clinical use | Three months
  After the standard folliculometry, will request the patient for self-performing scan (3D ultrasound)
Determination of the risks during use SMD | Three months
  Patients will have phone connection to call the nurse if any problems happen or when they finish the scan.

SECONDARY OUTCOMES:
Patient's perception as a user of the SMD | Three months
  To know the patient's perception as a user of the SMD by means of a satisfaction questionnaire
To recopilate the pelvic ultrasound volumes | Three months
  To recopilate the pelvic ultrasound volumes (uterus and ovaries inside) during COS exams for posterior development of an automated segmentation system (of the uterus and the ovaries) in the context of a next project, conditioned to the obtention of satisfactory outcomes after the finalization of the present study.

CONTACTS AND LOCATIONS:
Overall Officials: Marcos Ferrando Serrano, MD, Principal Investigator — IVI Bilbao; Pedro Royo Manero, Principal Investigator — IVI Bilbao
Locations (1):
- Ivi Bilbao, Bilbao, Bizkaia, Spain

IPD SHARING:
Plan to Share IPD: No